CLINICAL TRIAL: NCT05203367
Title: Randomized, Double-Blind, Placebo-Controlled, Phase 1 Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single-Ascending Doses of BAR 502 in Healthy Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BAR 502 in Healthy Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Update development program
Sponsor: BAR Pharmaceuticals s.r.l. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: BLCL-BAR-502-101
Record Dates: First submitted 2021-12-04; First posted 2022-01-24 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Non-alcoholic fatty liver disease; healthy; BAR 502
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — BAR502

STUDY DESIGN:
Intervention Model Description: A maximum of 4 BAR 502 dose levels are preplanned to be investigated in separate sequential cohorts. Each of these cohorts will consist of 8 healthy male and female subjects (3 subjects of either sex on active treatment, 1 of either sex on placebo).
  Each subject will participate in only one cohort.
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAR 502 (Experimental): Each subject will receive an oral single-dose of BAR 502.
  Interventions: Drug: BAR502
- Placebo (Placebo Comparator): Each subject will receive an oral single-dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAR502 — Single oral doses of BAR 502/placebo will be administered as film-coated tablets, in the morning of Day 1, with 240 mL of water, after an overnight fasting of at least 8 hours.
  BAR 502 film-coated tablets are available at dose strengths of 10, 50 and 150 mg. A maximum of 4 dose levels are pre-planned (10 mg, 50 mg, 150 mg, 300 mg).
  Arms: BAR 502
Drug: Placebo — Matching BAR 502 placebo film-coated tablets will be given to 2 out of 8 subjects in each cohort using the same regimen as outlined for the active study treatment
  Arms: Placebo

SUMMARY:
This is a prospective, single-center, randomized, double-blind, placebo-controlled, single-ascending dose (SAD) phase 1 study to evaluate the safety and tolerability of single-ascending doses of BAR 502 in healthy male and female subjects.

DETAILED DESCRIPTION:
This clinical trial will be the first-in-Human (FiH) study of BAR 502.

This study is planned to investigate up to 4 dose levels of BAR 502. Each dose level will consist of 8 healthy male and female subjects (ratio 1:1, male: female) to have 6 subjects being administered BAR 502 and 2 subjects being administered placebo (ratio 3:1, active: placebo).

The study is designed to meet the following objectives:

* Primary:

  * To evaluate the safety and tolerability of single-ascending doses of BAR 502 in healthy male and female subjects.
* Secondary:

  * To investigate the pharmacokinetics (PK) of single-ascending doses of BAR 502 in healthy male and female subjects;
  * To investigate the pharmacodynamics (PD) of single-ascending doses of BAR 502 in healthy male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent in a language understandable to the subject prior to any study-mandated procedure.
2. Ability to communicate well with the investigator, and to understand and comply with the study requirements.
3. Healthy male or female subject aged between 18 and 55 years (inclusive) at Screening.
4. Body mass index (BMI) of 18.0 to 30.0 kg/m2 (inclusive) at Screening.
5. Systolic blood pressure (SBP) 90-140 mmHg, diastolic blood pressure (DBP) 50-90 mmHg, and pulse rate 45-90 bpm (inclusive), measured on same arm after ≥5 min in the seated position, at Screening.
6. Estimated glomerular filtration rate calculated using the Cockcroft-Gault equation and normalized to an average surface area of 1.73 m2 ≥ 90 mL/min at Screening.
7. If woman, she meets one of the following criteria:

   1. is of non-childbearing potential; or
   2. is of childbearing potential and agrees to use an accepted non-hormonal or hormonal contraceptive method.

If man, he is infertile, vasectomized (i.e. who has received medical assessment of the surgical success) or agrees to abstain from or to use a condom during heterosexual intercourse with a woman of childbearing potential or a pregnant woman, and agrees not to donate sperm, from investigational product administration until at least 90 days after the investigational product administration. In addition, the subject must ensure that his female partner of childbearing potential agrees to consistently and correctly use one of the acceptable contraceptive methods mentioned above, for the same period of time.

Exclusion Criteria:

- At screening:

1. Previous exposure to BAR 502.
2. Known hypersensitivity to BAR 502, or any of its excipients.
3. Clinically relevant findings on physical examination.
4. Clinically relevant abnormalities on 12-lead ECG, measured after 5 min in a supine position.
5. Clinically relevant findings in clinical laboratory tests (hematology, clinical chemistry, and urinalysis).
6. QTcF > 450 ms in males and > 470 ms in females.
7. Medical history and/or clinical or laboratory evidence of liver or hepatobiliary disease or liver injury as indicated by serum alanine aminotransferase (ALT), AST, gamma-glutamyl transferase (GGT), ALP or total bilirubin levels exceeding the upper limit of normal (ULN).
8. International Normalized Ratio (INR) > 1.2.
9. Any medical condition, acute, ongoing, recurrent or chronic, that presents a potential risk to the participant and/or that may compromise the objectives of the study.
10. History of major medical or surgical disorders which, in the opinion of the investigator, are likely to interfere with the distribution, metabolism, or excretion of the investigational product.
11. History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to Screening.
12. Previous clinically relevant history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions.
13. Veins unsuitable for intravenous puncture on either arm (e.g., veins that are difficult to locate, access, or puncture, veins with a tendency to rupture during or after puncture).
14. Participation in a clinical study involving investigational product administration within 3 months prior to Screening or in more than 2 clinical studies within 1 year prior to Screening.
15. Excessive methylxanthines consumption, defined as ≥ 800 mg per day.
16. Nicotine intake (e.g., smoking, nicotine patch, nicotine chewing gum, or electronic cigarettes) within 3 months prior to Screening and inability to refrain from nicotine intake from Screening up to End-of-Study (EOS).
17. Loss of 250 mL or more of blood within 3 months prior to Screening.
18. Positive hepatitis B surface antigen (HBsAg) and/or hepatitis C virus antibodies.
19. Positive human immunodeficiency virus (HIV1 and HIV2) antibodies.
20. Positive results in urine drugs-of-abuse, cotinine or ethanol tests.
21. If woman, she is breastfeeding.
22. Positive result in serum pregnancy test.
23. Any other circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol or may render the subject unsuitable for the study.

    - At admission to treatment period:
24. Positive or inconclusive SARS-CoV-2 test result using polymerase chain reaction (PCR) technology prior to Admission to the clinical site.
25. Any recent disease or condition or treatment that, according to the Investigator, would put the subject at undue risk due to study participation or occurred at a timeframe in which may interfere with the study outcomes.
26. Clinically relevant findings on physical examination.
27. Clinically relevant abnormalities on 12-lead ECG, measured after 5 min in a supine position.
28. Clinically relevant findings in clinical laboratory tests.
29. Use of prescription or nonprescription medicinal products, including vitamins, food supplements, herbal supplements (including St John's Wort), within 3 weeks prior to study treatment administration, unless in the Investigator's opinion the medication does not interfere with the pharmacokinetics of study drug or compromise subject safety.
30. Consumption of Seville oranges, pomelo, pomegranate, starfruit or grapefruit products (fresh, canned, or frozen) since Screening.
31. Positive result in urine drugs-of-abuse, cotinine or ethanol tests.
32. Positive result in urine pregnancy test.
33. Any other condition that the investigator considers to render the subject unsuitable for the treatment period.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-25 (Estimated); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Through study completion, an average of 2 months
  Safety will be evaluated through the assessment of adverse events
Assessment of physical examination | At screening (Day -21 to Day -3 for male and female subjects of non-childbearing potential, Day -28 to Day -7 for female subjects of childbearing potential) and end of study ( Day 8)
  Safety will be evaluated through the assessment of physical examination, which will include: general appearance; skin; head and neck; thorax and abdomen; pulmonary auscultation; cardiac auscultation; abdomen palpation; limbs.
Assessment of 12-lead electrocardiogram | At screening (Day -21 to Day -3 for male and female subjects of non-childbearing potential, Day -28 to Day -7 for female subjects of childbearing potential), admission (Day-1), and from day 1 to day 4 of the study
  Safety will be evaluated through the assessment of 12-lead ECG. The following variables are to be collected on the eCRF: HR (bpm), and the intervals PR (ms), QRS (ms), QT (ms), QTcB (ms) and QTcF (ms).
Change from baseline at each time point of measurement in supine blood pressure (both systolic and diastolic) | At screening (Day -21 to Day -3 for male and female subjects of non-childbearing potential, Day -28 to Day -7 for female subjects of childbearing potential), admission (Day -1), from Day 1 to Day 4 of the study, and at end of study (at Day 8).
  Safety will be evaluated through the assessment of vital signs (systolic and diastolic blood pressure)
Change from baseline at each time point of measurement in pulse rate | At screening (Day -21 to Day -3 for male and female subjects of non-childbearing potential, Day -28 to Day -7 for female subjects of childbearing potential), admission (Day -1), from day 1 to day 4 of the study, and at end of study (at Day 8)..
  Safety will be evaluated through the assessment of vital signs

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | Within 1 hour prior to treatment administration and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 74 hours after treatment administration.
  Determination of BAR 502 concentrations in plasma, to investigate the pharmacokinetics
Time of occurrence of Cmax (Tmax) | Within 1 hour prior to treatment administration and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 74 hours after treatment administration.
  Determination of BAR 502 concentrations in plasma, to investigate the pharmacokinetics
Area under the plasma concentration-time curve (AUC) from time zero to last sampling time with quantifiable concentrations (AUC0-t); | Within 1 hour prior to treatment administration and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 74 hours after treatment administration.
  Determination of BAR 502 concentrations in plasma, to investigate the pharmacokinetics
AUC extrapolated to infinity | Within 1 hour prior to treatment administration and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 74 hours after treatment administration.
  Determination of BAR 502 concentrations in plasma, to investigate the pharmacokinetics
Apparent terminal elimination rate constant (λz); and apparent terminal elimination half-life (t1/2) | Within 1 hour prior to treatment administration and at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 74 hours after treatment administration.
  Determination of BAR 502 concentrations in plasma to investigate the pharmacokinetics
Cumulative amount of drug excreted in urine (AmtCUM) | From treatment administration to day 4 of the study
  Determination of BAR 502 concentrations in urine to investigate the pharmacokinetics
Area under the urine excretion curve (AUR) from time zero to last observed concentration (AURClast) | From treatment administration to day 4 of the study
  Determination of BAR 502 concentrations in urine to investigate the pharmacokinetics
Maximum rate of urinary excretion (Rmax) | From treatment administration to day 4 of the study
  Determination of BAR 502 concentrations in urine to investigate the pharmacokinetics
Percentage of drug recovered in urine (REC%) | From treatment administration to day 4 of the study
  Determination of BAR 502 concentrations in urine to investigate the pharmacokinetics
Time to Rmax (tumax) | From treatment administration to day 4 of the study
  Determination of BAR 502 concentrations in urine to investigate the pharmacokinetics
Renal clearance (CLR) | From treatment administration to day 4 of the study
  Determination of BAR 502 concentrations in urine to investigate the pharmacokinetics
Serum concentrations of total bile acids over time up to 24 hours post-dose | At admission, within 1 hour prior to study treatment administration, and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 16 and 24 hours after treatment administration.
  To investigate the pharmacodynamics
Serum concentrations of FGF19 over time up to 24 hours post-dose. | At admission, within 1 hour prior to study treatment administration, and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 16 and 24 hours after treatment administration
  To investigate the pharmacodynamics (biomarkers of Farnesoid X Receptor (FXR) target engagement)
Serum concentrations of C4 over time up to 24 hours post-dose. | At admission, within 1 hour prior to study treatment administration, and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 16 and 24 hours after treatment administration
  To investigate the pharmacodynamics (biomarkers of Farnesoid X Receptor (FXR) target engagement)
Serum concentrations of GLP-1 over time up to 24 hours post-dose. | At admission, within 1 hour prior to study treatment administration, and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 16 and 24 hours after treatment administration
  To investigate the pharmacodynamics (marker of G protein-coupled bile acid-activated receptor 1 (GPBAR1) activation)

CONTACTS AND LOCATIONS:
Locations (1):
- BlueClinical Phase I, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No